CLINICAL TRIAL: NCT02403076
Title: Management of Patients With Gastrointestinal Bleeding - a Prospective Single Center Registry Study
Brief Title: Gastrointestinal Bleeding Management
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: HSK006
Record Dates: First submitted 2015-03-12; First posted 2015-03-31 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
Unlike the management of patients with various forms of accidents (e.g. polytrauma), only a few data exists for the emergency management of patients with acute gastrointestinal bleeding. The aim of our study is to develop optimal diagnostic and therapeutic algorithms for the management of acute upper and lower gastrointestinal bleedings.

DETAILED DESCRIPTION:
Acute upper gastrointestinal bleeding is a common medical emergency. Up to 15% of patients still die worldwide. The gastroduodenal ulcer disease is the most common cause of gastrointestinal bleeding. Even lower gastrointestinal bleeding occurs especially in patients of older age.

The goal of our data acquisition and evaluation is to learn whether existing diagnostic or therapeutic procedures are of relevance in the management of acute gastrointestinal bleedings. Unlike the management of patients with various forms of accidents (e.g. polytrauma), only a few data exists on patients with acute gastrointestinal bleedings. The aim of our study is to develop optimal diagnostic and therapeutic algorithms of acute gastrointestinal bleeding. Therefore our prospective data registry should answer different questions:

When is the right time for a gastroscopy or colonoscopy? Should every patient with a suspected gastrointestinal bleeding receive endoscopy? Which clinical und laboratory findings influence the success of therapy? Does endoscopic procedures have an influence on the length of hospital stay?

Against this background we will record treatment findings separately. This includes clinical (e.g. age, sex, date of admission, department of admission, onset of symptoms), laboratory (e.g. blood count), history of medications (e.g. new anticoagulation's) and endoscopic findings (e.g. active bleeding). Furthermore the length of inhospital stay will be recorded.

Participants will be followed for the duration of hospital stay, an expected average of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* All patients with suspicion or symptoms of gastrointestinal bleeding.

Exclusion Criteria:

* Patients younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients that will be admitted to our hospital with a gastrointestinal bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Time of endoscopy | Participants will be followed for the duration of hospital stay, an expected average of 7 days.
  The aim of this primary endpoint should reflect whether the timing of endoscopic diagnosis after admission has an impact on the length hospital stay.

SECONDARY OUTCOMES:
Follow up endoscopy (how many patients with gastrointestinal bleeding receive follow-up endoscopy ) | Participants will be followed for the duration of hospital stay, an expected average of 7 days.
  It will be noted how many patients with gastrointestinal bleeding receive follow-up endoscopy with therapeutic procedures.
Endoscopic therapies (whether taking anticoagulants have an impact on the need for endoscopic therapies) | Participants will be followed for the duration of hospital stay, an expected average of 7 days.
  It should be study whether taking anticoagulants have an impact on the need for endoscopic therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kiesslich, Professor, Study Director — HSK Clinic Wiesbaden, Department of Internal Medicine II